CLINICAL TRIAL: NCT02771808
Title: Haptoglobin Polymorphism as a Determinant of Adverse Outcome After Cardiac Surgery in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: International Anesthesia Research Society (IARS) (Other)
Responsible Party: Principal Investigator, Jacob Raphael, Associate Professor of Anesthesiology, University of Virginia
Other Study IDs: 14691
Record Dates: First submitted 2010-09-17; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Artery Disease
Keywords: CABG
MeSH Terms: conditions — Coronary Artery Disease | interventions — Haptoglobins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diabetic patients: obtain biomarker samples from diabetic patients and examine for 1-1 & 1-2 & 2-2 haptoglobin genotype
  Interventions: Other: biomarker samples

INTERVENTIONS:
Other: biomarker samples — biomarker samples for haptoglobin genotype (RT-PCR) and phenotype (hemoglobin electrophoresis) general markers for oxidative stress (isoprostane f2 alpha, malondialdehyde) markers of inflammation (CRP, IL-1, 2, 6, 10 and TNF) markers of cardiac injury (CPK, troponins and BNP) markers of kidney injury (cystatin C, creatinine, GFR)
  Other Names: haptoglobin

SUMMARY:
Specific aim 1a will test the hypothesis that diabetic patients with 2-2 haptoglobin genotype have higher indices of postoperative myocardial injury (creatine kinase MB isoenzyme , Troponin I ) and renal injury (as indicated by elevated creatinine, cytostatin C and glomerular filtration rate). Of note, significantly elevated levels (>5 times the upper normal limit) of creatine kinase MB isoenzyme and troponins postoperatively have been associated with postoperative myocardial ischemia/infarction and are a predictor of short-term and long-term mortality after cardiac surgery.

Specific aim 1b will evaluate preoperative and postoperative indices of oxidative stress (such as isoprostane f2 alpha and malondialdehyde) and will evaluate whether patients with type 2-2 haptoglobin express increased oxidative stress. The investigators will also try to correlate whether patients with increased oxidative stress are those with elevated indices of myocardial and/or renal injury Specific aim 1c will try to evaluate whether patients with type 2-2 haptoglobin also have increased levels of inflammatory indices (C-reactive protein,[interleukin] IL-1, IL-2, IL-6, TNF[tumor necrosis factor]) and try to correlate the findings with postoperative myocardial and or renal injury.

The incidence of atrial fibrillation after coronary artery bypass graft ranges from 19% to 27%. The investigators will also look at any correlation of the type 2-2 haptoglobin and the incidence of post-operative atrial fibrillation.

DETAILED DESCRIPTION:
Diabetes mellitus is a major risk factor for postoperative morbidity and mortality after cardiac surgery, mainly because of accelerated atherosclerosis and target-organ injury that predispose these patients to increased incidence of postoperative morbidity (such as but not limited to, postoperative adverse cardiac events, renal injury or stroke) and mortality.

Over the past several years haptoglobin has been identified as a risk factor that predicts the development of cardiovascular complications in diabetics. There are 3 major haplotypes of haptoglobin: 1-1; 1-2 and 2-2. Several studies have demonstrated that diabetic individuals with the 2-2 genotype have up to 5 fold increased risk to develop cardiovascular complications as compared to diabetic patients with a non-2-2 haptoglobin genotype. There is no data in the literature that evaluated whether the haptoglobin 2-2 genotype is a risk factor for increased postoperative morbidity and/or mortality after cardiac surgery in patients with DM.

Therefore, the aims of the study are to evaluate whether diabetic patients with the 2-2 genotype are at increased risk for postoperative morbidity and/or mortality after cardiac surgery.

Preliminary studies in diabetic patients demonstrated that those with haptoglobin 2-2 genotype are at increased risk for cardiovascular complications of diabetes. Moreover, these patients were found to have increased in-hospital mortality after acute MI compared to diabetic individuals that do not have the 2-2 genotype, and they also suffer from increased incidence of post catheterization stent thrombosis compared to diabetics that do not have the 2-2 genotype

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Scheduled for an elective cardiac surgery on pump
* Diabetic -type I or type II
* Informed consent

Exclusion Criteria:

* Patients with chronic hemolytic disorders;
* Patients with hemoglobinopathies
* Enrollment in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult diabetic patients scheduled for an elective cardiac surgery on pump at UVA
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2010-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
number of participants with myocardial injury | 24 hours post CPB
  number of participants with general markers for myocardial injury

SECONDARY OUTCOMES:
number of participants with renal injury | 24 hrs post CPB
  number of participants with markers of kidney injury (cystatin C, creatinine, GFR)
number of participants with incidence of new onset atrial fibrillation | day 15
  incidence of new onset atrial fibrillation will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Raphael, MD, Principal Investigator — UVA Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno PR, Fuster V. New aspects in the pathogenesis of diabetic atherothrombosis. J Am Coll Cardiol. 2004 Dec 21;44(12):2293-300. doi: 10.1016/j.jacc.2004.07.060. PMID 15607389
- [Background] Donahoe SM, Stewart GC, McCabe CH, Mohanavelu S, Murphy SA, Cannon CP, Antman EM. Diabetes and mortality following acute coronary syndromes. JAMA. 2007 Aug 15;298(7):765-75. doi: 10.1001/jama.298.7.765. PMID 17699010
- [Background] Bucerius J, Gummert JF, Walther T, Doll N, Falk V, Onnasch JF, Barten MJ, Mohr FW. Impact of diabetes mellitus on cardiac surgery outcome. Thorac Cardiovasc Surg. 2003 Feb;51(1):11-6. doi: 10.1055/s-2003-37280. PMID 12587082
- [Background] Carson JL, Scholz PM, Chen AY, Peterson ED, Gold J, Schneider SH. Diabetes mellitus increases short-term mortality and morbidity in patients undergoing coronary artery bypass graft surgery. J Am Coll Cardiol. 2002 Aug 7;40(3):418-23. doi: 10.1016/s0735-1097(02)01969-1. PMID 12142105
- [Background] Thourani VH, Weintraub WS, Stein B, Gebhart SS, Craver JM, Jones EL, Guyton RA. Influence of diabetes mellitus on early and late outcome after coronary artery bypass grafting. Ann Thorac Surg. 1999 Apr;67(4):1045-52. doi: 10.1016/s0003-4975(99)00143-5. PMID 10320249
- [Background] Levy AP, Hochberg I, Jablonski K, Resnick HE, Lee ET, Best L, Howard BV; Strong Heart Study. Haptoglobin phenotype is an independent risk factor for cardiovascular disease in individuals with diabetes: The Strong Heart Study. J Am Coll Cardiol. 2002 Dec 4;40(11):1984-90. doi: 10.1016/s0735-1097(02)02534-2. PMID 12475459
- [Background] Roguin A, Koch W, Kastrati A, Aronson D, Schomig A, Levy AP. Haptoglobin genotype is predictive of major adverse cardiac events in the 1-year period after percutaneous transluminal coronary angioplasty in individuals with diabetes. Diabetes Care. 2003 Sep;26(9):2628-31. doi: 10.2337/diacare.26.9.2628. PMID 12941730
- [Background] Suleiman M, Aronson D, Asleh R, Kapeliovich MR, Roguin A, Meisel SR, Shochat M, Sulieman A, Reisner SA, Markiewicz W, Hammerman H, Lotan R, Levy NS, Levy AP. Haptoglobin polymorphism predicts 30-day mortality and heart failure in patients with diabetes and acute myocardial infarction. Diabetes. 2005 Sep;54(9):2802-6. doi: 10.2337/diabetes.54.9.2802. PMID 16123372
- [Background] Asleh R, Guetta J, Kalet-Litman S, Miller-Lotan R, Levy AP. Haptoglobin genotype- and diabetes-dependent differences in iron-mediated oxidative stress in vitro and in vivo. Circ Res. 2005 Mar 4;96(4):435-41. doi: 10.1161/01.RES.0000156653.05853.b9. Epub 2005 Jan 20. PMID 15662028
- [Background] Guetta J, Strauss M, Levy NS, Fahoum L, Levy AP. Haptoglobin genotype modulates the balance of Th1/Th2 cytokines produced by macrophages exposed to free hemoglobin. Atherosclerosis. 2007 Mar;191(1):48-53. doi: 10.1016/j.atherosclerosis.2006.04.032. Epub 2006 Jul 3. PMID 16820150
- [Background] Greenson N, Macoviak J, Krishnaswamy P, Morrisey R, James C, Clopton P, Fitzgerald R, Maisel AS. Usefulness of cardiac troponin I in patients undergoing open heart surgery. Am Heart J. 2001 Mar;141(3):447-55. doi: 10.1067/mhj.2001.113071. PMID 11231444
- [Background] Muehlschlegel JD, Perry TE, Liu KY, Nascimben L, Fox AA, Collard CD, Avery EG, Aranki SF, D'Ambra MN, Shernan SK, Body SC; CABG Genomics Investigators. Troponin is superior to electrocardiogram and creatinine kinase MB for predicting clinically significant myocardial injury after coronary artery bypass grafting. Eur Heart J. 2009 Jul;30(13):1574-83. doi: 10.1093/eurheartj/ehp134. Epub 2009 Apr 30. PMID 19406870
- [Background] Paparella D, Cappabianca G, Visicchio G, Galeone A, Marzovillo A, Gallo N, Memmola C, Schinosa Lde L. Cardiac troponin I release after coronary artery bypass grafting operation: effects on operative and midterm survival. Ann Thorac Surg. 2005 Nov;80(5):1758-64. doi: 10.1016/j.athoracsur.2005.04.040. PMID 16242452
- [Background] Ramsay J, Shernan S, Fitch J, Finnegan P, Todaro T, Filloon T, Nussmeier NA. Increased creatine kinase MB level predicts postoperative mortality after cardiac surgery independent of new Q waves. J Thorac Cardiovasc Surg. 2005 Feb;129(2):300-6. doi: 10.1016/j.jtcvs.2004.06.005. PMID 15678039
- [Background] Adabag AS, Rector T, Mithani S, Harmala J, Ward HB, Kelly RF, Nguyen JT, McFalls EO, Bloomfield HE. Prognostic significance of elevated cardiac troponin I after heart surgery. Ann Thorac Surg. 2007 May;83(5):1744-50. doi: 10.1016/j.athoracsur.2006.12.049. PMID 17462392
- [Background] Fox AA, Shernan SK, Collard CD, Liu KY, Aranki SF, DeSantis SM, Jarolim P, Body SC. Preoperative B-type natriuretic peptide is as independent predictor of ventricular dysfunction and mortality after primary coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2008 Aug;136(2):452-61. doi: 10.1016/j.jtcvs.2007.12.036. PMID 18692657
- [Background] Cuthbertson BH, Croal BL, Rae D, Gibson PH, McNeilly JD, Jeffrey RR, Smith WC, Prescott GJ, Buchan KG, El-Shafei H, Gibson GA, Hillis GS. N-terminal pro-B-type natriuretic peptide levels and early outcome after cardiac surgery: a prospective cohort study. Br J Anaesth. 2009 Nov;103(5):647-53. doi: 10.1093/bja/aep234. Epub 2009 Aug 27. PMID 19713279
- [Background] Bahar I, Akgul A, Ozatik MA, Vural KM, Demirbag AE, Boran M, Tasdemir O. Acute renal failure following open heart surgery: risk factors and prognosis. Perfusion. 2005 Oct;20(6):317-22. doi: 10.1191/0267659105pf829oa. PMID 16363316
- [Background] Brown JR, Cochran RP, Leavitt BJ, Dacey LJ, Ross CS, MacKenzie TA, Kunzelman KS, Kramer RS, Hernandez F Jr, Helm RE, Westbrook BM, Dunton RF, Malenka DJ, O'Connor GT; Northern New England Cardiovascular Disease Study Group. Multivariable prediction of renal insufficiency developing after cardiac surgery. Circulation. 2007 Sep 11;116(11 Suppl):I139-43. doi: 10.1161/CIRCULATIONAHA.106.677070. PMID 17846294
- [Background] McGuinness J, Bouchier-Hayes D, Redmond JM. Understanding the inflammatory response to cardiac surgery. Surgeon. 2008 Jun;6(3):162-71. doi: 10.1016/s1479-666x(08)80113-8. PMID 18581753
- [Background] Warren OJ, Smith AJ, Alexiou C, Rogers PL, Jawad N, Vincent C, Darzi AW, Athanasiou T. The inflammatory response to cardiopulmonary bypass: part 1--mechanisms of pathogenesis. J Cardiothorac Vasc Anesth. 2009 Apr;23(2):223-31. doi: 10.1053/j.jvca.2008.08.007. Epub 2008 Oct 19. No abstract available. PMID 18930659
- [Background] Paparella D, Yau TM, Young E. Cardiopulmonary bypass induced inflammation: pathophysiology and treatment. An update. Eur J Cardiothorac Surg. 2002 Feb;21(2):232-44. doi: 10.1016/s1010-7940(01)01099-5. PMID 11825729
- [Background] Orhan G, Yapici N, Yuksel M, Sargin M, Senay S, Yalcin AS, Aykac Z, Aka SA. Effects of N-acetylcysteine on myocardial ischemia-reperfusion injury in bypass surgery. Heart Vessels. 2006 Jan;21(1):42-7. doi: 10.1007/s00380-005-0873-1. PMID 16440148